CLINICAL TRIAL: NCT01475799
Title: Evaluation of the Direct Flow Medical Percutaneous Aortic Valve 18F System for the Treatment of Patients With Severe Aortic Stenosis
Brief Title: Percutaneous Aortic Valve 18F System for the Treatment of Patients With Severe Aortic Stenosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Direct Flow Medical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IP 010
Record Dates: First submitted 2011-11-17; First posted 2011-11-21 (Estimated); Last update posted 2016-11-01 (Estimated); Status verified 2016-10

CONDITIONS: Aortic Valve Stenosis
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Percutaneous Aortic Valve 18F System (Experimental): Evaluation of the Direct Flow Medical Percutaneous Aortic Valve 18F System for the Treatment of Patients with Severe Aortic Stenosis.
  Interventions: Device: Replacement of the Aortic Stenotic Valve

INTERVENTIONS:
Device: Replacement of the Aortic Stenotic Valve — Treatment for patients with Severe Aortic Stenosis.
  Other Names: TAVR

SUMMARY:
The purpose of the study is to determine the safety and performance of the Direct Flow Medical study valve and delivery procedure.

DETAILED DESCRIPTION:
Prospective, multicenter, non-randomized clinical trial of the Direct Flow Medical Percutaneous Aortic Valve 18F System for the treatment of severe aortic stenosis

ELIGIBILITY:
Inclusion Criteria

All candidates for the study must meet the following inclusion criteria:

1. Severe aortic valve stenosis determined by echocardiogram and Doppler, defined as: mean gradient >40 mmHg or peak jet velocity >4.0 m/s and an aortic valve area ≤0.8 cm2 or aortic valve area index ≤0.5 cm2/m2
2. Symptomatic aortic valve stenosis demonstrated by angina, congestive heart failure, NYHA Functional Class ≥ II, or syncope
3. Patient is an extreme risk candidate for open surgical aortic valve repair such that the site Investigators (interventional cardiologist and cardiothoracic surgeon) agree that medical factors preclude operation, based on the conclusion that the probability of death or serious morbidity exceeds the probability of meaningful improvement due to the patient's co-morbidities (such as, but not limited to, severe COPD, porcelain aorta, previous thorax irradiation) or logistic EuroSCORE ≥ 20
4. ≥ 70 years old
5. Patient has been informed of the nature of the study and has provided written informed consent
6. Patient and treating physician agree that the patient will return for all required post-procedure follow-up visits

Exclusion Criteria

Candidates will be excluded from the study if any of the following criteria are present:

1. Patient is a surgical candidate for aortic valve replacement
2. Congenital bicuspid or unicuspid valve determined by echocardiography
3. Native valve annulus diameter is <17mm or >22mm determined by the screening CT scan
4. Extreme asymmetrical calcification of the native aortic valve determined by the screening CT scan
5. Native valvular or peripheral vascular anatomy is not appropriate for the DFM bioprosthesis and 18F delivery system
6. Left ventricular ejection fraction (LVEF) <30% determined by resting echocardiogram
7. Evidence of an acute myocardial infarction (Refer to Definitions in Section 8) within 30 days prior to the study procedure
8. Any percutaneous coronary or peripheral interventional procedure performed within 30 days prior to the study procedure
9. Any planned surgical or percutaneous coronary or peripheral procedure to be performed during the study procedure or prior to 30 day follow-up visit
10. Need for emergency surgery for any reason
11. Untreated clinically significant ( > 70% obstruction) coronary artery disease requiring revascularization
12. Prior aortic or mitral valve surgery
13. Pre-existing prosthetic heart valve in any position
14. Mitral insufficiency greater than moderate determined by resting echocardiography
15. Echocardiographic evidence of intra-cardiac mass, thrombus or vegetation
16. Thoracic aortic aneurysm (TAA)
17. Abdominal aortic aneurysm (AAA) >4.5 cm
18. Presence of an endovascular stent graft for treatment of AAA or TAA
19. Hypertrophic cardiomyopathy
20. Hemodynamic instability (e.g. requiring inotropic support)
21. Trans-esophageal echocardiography (TEE) is contraindicated
22. Renal insufficiency (creatinine > 3.0 mg/dL) and/or end-stage renal disease requiring dialysis at the time of screening
23. Active endocarditis or sepsis within 6 months prior to the study procedure
24. Stroke or transient ischemic attack (TIA) within 6 months prior to the study procedure
25. Cardiogenic shock within 30 days prior to the study procedure
26. Active peptic ulcer or upper GI bleeding within 3 months prior to the study procedure
27. Leukopenia (WBC <3000/mm³), acute anemia (Hb <9 g/dL), or thrombocytopenia (platelet count <100,000 cells/mm3)
28. History of bleeding diathesis or coagulopathy or refusal of blood transfusions
29. A known hypersensitivity or contraindication to aspirin, heparin, ticlopidine or clopidogrel, or sensitivity to contrast media, which cannot be adequately pre-medicated
30. Currently participating in an investigational drug or another device trial
31. Previously enrolled in this study
32. Patient refusal of surgery
33. Life expectancy thought to be <12 months
34. Dementia (resulting in either inability to provide informed consent for the trial/procedure, prevents independent lifestyle outside of a chronic care facility, or will fundamentally complicate rehabilitation from the procedure or compliance with follow-up visits)

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 112 (Actual)
Dates: Start 2011-11; Primary Completion 2014-07 (Actual); Study Completion 2019-07 (Estimated)

PRIMARY OUTCOMES:
Freedom from all-cause mortality from procedure to 30 days | Procedure to 30 days

SECONDARY OUTCOMES:
Device Success at procedure completion | At procedure completion
  Device success is assessed at the completion of the study procedure based on TEE

CONTACTS AND LOCATIONS:
Overall Officials: Thierry LeFevre, M.D., Principal Investigator — Study PI; Prof. Joachim Schofer, Principal Investigator — Study PI
Locations (12):
- France (2):
  - L'Institut Hospitalier Jacques Cartier, Massy
  - Clinique Pasteur, Toulouse
- Germany (5):
  - Vivantes Klinikum im Friedrichshain, Berlin, DE
  - University Hospital Bonn, Bonn
  - Elisabeth-Krankenhaus Essen, GmbH, Essen
  - Medical Care Center, Prof Mathey, Prof Schofer, Hamburg
  - Krankenhaus der Barmherzigen Brüder Trier, Trier
- Italy (2):
  - San Raffaele Hospital, Milan
  - Azienda Ospedaliera Niguarda Ca Granda, Milan
- Centre hospitalier de Luxembourg, Luxembourg, Luxembourg
- United Kingdom (2):
  - St. Thomas' Hospital, London, London
  - St. Bartholomew's Hospital, London